CLINICAL TRIAL: NCT06632145
Title: Cog-Fun Ageing Participation-centered, Health Promotion for Older Adult
Brief Title: Cog-Fun Ageing Participation-centered, Health Promotion for Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, Adina Maeir, Prof. Adina Maeir, School of Occupational Therapy Hebrew University, Hebrew University of Jerusalem
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 04042023
Record Dates: First submitted 2024-10-06; First posted 2024-10-08 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Subjective Cognitive Decline (SCD)
Keywords: Occupational experience; Participation; Cognitive functional interventions; Functional decline

STUDY DESIGN:
Intervention Model Description: Pre post pilot feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cog Fun Ageing intervention (Experimental)
  Interventions: Other: Cog Fun Ageing intervention

INTERVENTIONS:
Other: Cog Fun Ageing intervention — Cog Fun Ageing is a group-based occupation-centered intervention aimed at promoting positive occupational experiences despite cognitive challenges in day to day life. The intervention includes 14 weekly 120-minute group sessions led by experienced occupational therapists. Sessions incorporate learning about the bio-psycho-social factors of SCD and strategies to manage and cope with occupational challenges resulting from SCD.

SUMMARY:
The goal of this feasibility study is to test the feasibility of a group intervention program based on health management principles for older adults with Subjective Cognitive Decline (SCD). SCD is a condition where individuals feel that their memory is worsening, although standard tests do not detect it. This perceived memory decline can lead to negative feelings and self-perception, causing people to withdraw from meaningful activities.

This study aims to answer three main questions:

1. Is the intervention feasible in terms of fidelity, adherence, and participant satisfaction?
2. Are the assessments used sensitive enough to identify the unique challenges faced by the SCD population and detect changes after the intervention?
3. What are the preliminary effects of the intervention on participants' perceptions of how SCD affects their daily life, mental health, and quality of life?

Participants will:

1. Take part in 14 weekly group sessions focused on managing the challenges of living with SCD and improving participation in daily activities.
2. Complete assessments before and after the intervention to measure their satisfaction with the program, and track changes in their perceptions of daily life, mental health, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported memory changes,
* A score of 23 or higher on the Montreal Cognitive Assessment (MoCA)
* Proficiency in Hebrew to participate fully in a Hebrew-speaking group.

Exclusion Criteria:

* Presence of a significant health condition that affects functioning
* Residence in a medical institution or nursing home
* Current participation in another SCD treatment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Memory Impact Questionnaire (MIQ) | After enrollment (before intervention) and 14 weeks later (after intervention)
  The Memory Impact Questionnaire (MIQ) will be used to assess the impact of perceived memory changes on daily life. The questionnaire was developed for use in both clinical and research settings to better understand the impact of memory changes on the day-to-day functioning of older adults and to monitor outcomes of support programs for this population. The questionnaire includes 51-item comprised of three subscales: Lifestyle Restrictions (19 items exploring social relationships, work, volunteer and leisure activities), Positive Coping (19 items exploring participation in cognitively engaging tasks and other positive responses to memory changes), and Negative Emotions (13 items exploring negative self-perceptions and perceived negative judgments from others). The total score, calculated by reverse-coding Positive Coping items and summing all items, reflects the overall burden of memory changes, with higher scores indicating a greater negative impact.

SECONDARY OUTCOMES:
Patient Health Questionnaire -4 (PHQ-4 ) | After enrollment (before intervention) and 14 weeks later (after intervention)
  The Patient Health Questionnaire-4 (PHQ-4) is a brief, self-report screening tool designed to quickly assess symptoms of depression and anxiety in the general population. It includes four questions, with two focused on anxiety and two on depression. The PHQ-4 combines two well-established scales: the PHQ-2 (depression) and the GAD-2 (anxiety).
  Participants respond to each question based on how often they have experienced certain symptoms over the past two weeks, using a 4-point Likert scale from 0 = Not at all to 3 = Nearly every day. The total score ranges from 0 to 12, with subscale scores ranging from 0 to 6 for both anxiety and depression. Scores are rated as: 0-2- Normal; 3-5 -Mild; 6-8- Moderate; 9-12- Severe.
  Total score ≥3 for first 2 questions suggests anxiety. Total score ≥3 for last 2 questions suggests depression.
SHARE version of the CASP-12 | After enrollment (before intervention) and 14 weeks later (after intervention)
  The CASP-12 (Control, Autonomy, Self-realization, and Pleasure) is a self-report questionnaire designed to measure the quality of life (QoL) in older adults, specifically targeting individuals aged 50 and over. The CASP-12 includes 12 items spread across four dimensions: control (the ability to influence one's environment), autonomy (freedom from external influence), self-realization (personal fulfillment), and pleasure (enjoyment in life).
  Participants rate each item on a 4-point Likert scale, ranging from 1 (often) to 4 (never), with higher scores indicating a higher quality of life. The total score can range from 12 to 48, where higher scores suggest greater well-being and satisfaction in the participants' lives.
Engagement in Meaningful Activities Survey (EMAS) | After enrollment (before intervention) and 14 weeks later (after intervention)
  The Engagement in Meaningful Activities Survey (EMAS) is a 12-item self-report questionnaire used to assess how meaningful a person's daily activities are. The survey asks participants to rate statements like "The activities I do give me a sense of satisfaction"; or "The activities I do help me feel competent," using a 4-point scale where 1 means "rarely"; and 4 means "always". The total score ranges from 12 to 48, with higher scores indicating higher levels of engagement in meaningful activities.
  This tool is used to measure changes in how participants perceive the value and meaning of their activities. The EMAS helps identify whether interventions improve participants' sense of purpose and satisfaction in their daily lives.

CONTACTS AND LOCATIONS:
Overall Officials: Adina Maeir, PhD, Principal Investigator — School of occupational therapy, faculty of medicine, Hebrew University
Locations (1):
- Hebrew University of Jerusalem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Due to the preliminary nature of the study, the outcome measures are still being evaluated for their suitability for interventions for the target population.

REFERENCES:
- [Background] Roheger M, Hennersdorf XS, Riemann S, Floel A, Meinzer M. A systematic review and network meta-analysis of interventions for subjective cognitive decline. Alzheimers Dement (N Y). 2021 Jul 12;7(1):e12180. doi: 10.1002/trc2.12180. eCollection 2021. PMID 34268448
- [Background] Rotenberg S, Leung C, Quach H, Anderson ND, Dawson DR. Occupational performance issues in older adults with subjective cognitive decline. Disabil Rehabil. 2022 Aug;44(17):4681-4688. doi: 10.1080/09638288.2021.1916626. Epub 2021 May 14. PMID 33989108